CLINICAL TRIAL: NCT02483390
Title: Use of Online Communications to Support Patients and Their Families in the Hospice Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pesach Shvartzman (Other)
Responsible Party: Sponsor-Investigator, Pesach Shvartzman, Prof., Meir Medical Center
Organization: Meir Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ק007/2015
Record Dates: First submitted 2015-06-10; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Palliative Care
Keywords: palliative care; e-health; e-therapy; psychosocial services
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group: All dyads are in the intervention arm. (Experimental)
  Interventions: Other: psychosocial intervention

INTERVENTIONS:
Other: psychosocial intervention — e-health services (e.g. by use of SKYPE) to the psychosocial needs of patients and their families who are getting services through home hospice care. In addition, the attitudes of the hospice staff will be investigated to the use of e-health methods.

SUMMARY:
The increasing awareness of the importance of palliative care has led, in Israel, to the 2005 Law for the Rights of Persons with Terminal Illness. Still, problems of accessibility to palliative care remain unresolved. The use of e-health services is likely to expand the ability of the medical, psychosocial and nursing staff to reach patients who are either living in the periphery, are unable to make clinic visits or whose family members are housebound in order to be caregivers. This exploratory research is designed to explore the issues, barriers and advantages of e-health care through the perspective of the palliative care staff members, the patients themselves and their caregiving family members.

DETAILED DESCRIPTION:
This study is designed to test the applicability and suitability of e-health services (e.g. by use of SKYPE) to the psychosocial needs of patients and their families who are getting services through home hospice care. In addition, the attitudes of the hospice staff will be investigated to the use of e-health methods. The study will clarify selection criteria, referral pathways and barriers and/or supporting elements that will allow e-health services to be provided in a highly professional fashion. Up to 20 dyads of a patient and their primary caregiver will be recruited from those who are receiving services from the home hospice unit of the Kupat Holim Clalit (General Sick Fund) in the South of Israel.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently receiving care from the home hospice unit,
* over the age of 18,
* able to give informed consent,
* with a computer that can use SKYPE or a smartphone,
* speaking a language of the psychosocial staff person (Hebrew, English, Russian, Arabic).

Exclusion Criteria:

* Brain tumors,
* dementia,
* speech disturbance,
* refusal to participate,
* language other than the four spoken by psychosocial staff members,
* inability to use technology or lack of computer in the home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
SWAT - The social work assessment tool | One year
  Tool to assess the quality of social work psychosocial services

SECONDARY OUTCOMES:
EIS (Emotional Intimacy Scale) | 6 month
  assess the emotional intimacy component a close relationship
SLDS (Satisfaction with cancer scale) | 6 month
  assess cancer patient quality of life
the will to live question | 6 month
  assess the will to live in a specific time point
ZBI (Zarit burden scale), | 6 month
  assess primary care burden
attitudes toward use of e-therapy questionnaire. | 6 month
  estimate attitudes of professional care giver